CLINICAL TRIAL: NCT04181879
Title: A Pilot Cluster Randomised Controlled Trial of a Theory-based Intervention to Improve Appropriate Polypharmacy in Older People in Primary Care
Brief Title: Appropriate Polypharmacy in Older People in Primary Care
Acronym: PolyPrime
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen's University, Belfast (Other)
Collaborators: University of Dublin, Trinity College (Other); Royal College of Surgeons, Ireland (Other); National University of Ireland, Galway, Ireland (Other); Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Carmel Hughes, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: B19/20
Record Dates: First submitted 2019-11-25; First posted 2019-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Polypharmacy
Keywords: Older people; Primary care; General Practitioners; Behaviour Change Techniques
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: A pilot cluster randomised controlled trial (cRCT). Eligible GP practices will be allocated to intervention or control (usual care) arm by a Northern Ireland Clinical Trials Unit (NICTU) statistician using an automated randomisation system. Practices will be randomised on a 1:1 allocation ratio stratified by country (i.e. Northern Ireland or the Republic of Ireland).
Who Masked: Outcomes Assessor
Masking Description: Members of the research team who are pharmacists will undertake an assessment of medication appropriateness following medication review by GPs and will be blind to the allocation of patients to either arm.
  Due to the nature of the intervention package (i.e. access to the video and patient recall), we will be unable to blind the GPs or patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): GPs will receive the intervention package and conduct medication reviews with recruited patients
  Interventions: Behavioral: Intervention
- Usual care (No Intervention): GPs will continue to treat recruited patients as usual

INTERVENTIONS:
Behavioral: Intervention — * GPs allocated to the intervention will be given access to the intervention package and asked to perform medication reviews with approximately 10 patients on two occasions (initial and 6-months follow-up).
  * The intervention package consists of two components: (a) an online video demonstrating how GPs can improve appropriate polypharmacy during typical consultations with older patients; (b) a patient recall process (appointment with the GP for a medication review).
  * GPs will be asked to schedule appointments with consenting patients (telephone or online consultations where a face-to-face consultation is not possible). During these appointments, GPs will undertake medication reviews ('a structured, critical examination of a person's medicines with the objective of reaching an agreement with the person about treatment, optimising the impact of medicines, minimising the number of medication-related problems and reducing waste').
  Other Names: PolyPrime
  Arms: Intervention

SUMMARY:
In the past, prescribing many medicines (polypharmacy) was seen in a negative light. However, because people are living longer and have several medical conditions at the same time, views on polypharmacy have changed. The challenge is to have the correct balance between enough medicines and too many medicines. Members of the research team have developed a new approach to achieving this balance. This approach has been tested in two general practices in Northern Ireland (NI). The approach (intervention package) currently consists of two parts: (1) a video showing how general practitioners (GPs) can prescribe appropriate polypharmacy for older patients, and (2) an appointment system for patients to visit a GP to have their medicines reviewed. As the intervention package was developed and tested in NI, further testing needs to be carried out in NI and the six border counties of the Republic of Ireland (ROI; Cavan, Donegal, Leitrim, Louth, Monaghan, and Sligo). This will be done in three stages or phases. In phase 1, which is now complete, 13 GPs were interviewed across 12 practices in the six border counties in the ROI; shown the video, asked about this new approach and asked if any changes are needed before doing more testing. In the next two phases (Phase 2 & 3) a small study will be carried out involving 12 practices: six practices in NI and six practices in the six border counties in the ROI and approximately 10 patients per practice. GP practices will either receive the intervention package and conduct medication reviews with recruited patients (intervention group) or continue to treat recruited patients as usual (control group). Interviews with up to 10 GPs and six members of practice staff (i.e. those involved in implementing the intervention within each practice) respectively in the six intervention group practices will also be conducted at the end of the intervention. Patients from the six intervention group practices will be asked to complete a feedback questionnaire after the delivery of the intervention (i.e. after completion of their final follow-up questionnaires).

DETAILED DESCRIPTION:
Design: We will perform a pilot cluster randomised controlled trial where 12 GP practices will be randomly assigned (6 GP practices per arm) to the intervention group versus usual care. Randomisation will be stratified according to location (Northern Ireland /Republic of Ireland - Cavan, Donegal, Leitrim, Louth, Monaghan and Sligo). GP practices will be randomly allocated to the intervention or usual care arm after patient screening and recruitment. A total of 120 patients (60 per study arm, approximately 10 patients, randomly selected, per GP practice) will be enrolled into the study.

Design: Pilot cluster randomized controlled trial

Unit of randomization: GP practice.

Unit of analysis: Patient and GP practice.

Setting: Practices located in Northern Ireland will be recruited via Research Nurse(s) from the Northern Ireland Clinical Research Network (NICRN - Primary Care). In the Republic of Ireland a Research Nurse(s) from Trinity College Dublin will recruit GP practices located in the border counties of Cavan, Donegal, Leitrim, Louth, Monaghan and Sligo.

Study aim: The overall aim of the study is to undertake a pilot cluster randomised controlled trial (cRCT) of a theory-based intervention targeting prescribing of appropriate polypharmacy in primary care (PolyPrime) to assess the feasibility of a definitive cRCT of the PolyPrime intervention.

The main study objectives are:

* To test approaches to sampling, recruitment and retention of GP practices
* To test approaches to screening, recruitment and retention of patients
* To test the feasibility of using medication appropriateness (assessed using the STOPP/START criteria) as the primary outcome in a future cRCT
* To identify the intervention's likely mechanism of action
* To assess if the intervention was delivered and received as intended (intervention fidelity)
* To identify the resources used in the set-up and delivery of the intervention and their associated costs
* To assess the feasibility of a future cost-effectiveness analysis
* To further validate the Medication-Related Burden quality of life (MRQ-QoL) tool
* To obtain estimates of effect size between groups, cluster size and intraclass correlation coefficients (ICCs) to inform the sample size calculation for a full RCT

Recruitment strategy for patients: Each recruited general practice will be asked to recruit 10 older patients meeting the inclusion criteria (i.e. over 70 years old, receiving four or more regular medicines, not cognitively impaired, not have a terminal illness, resident in the community, be in receipt of a valid general medical services (GMS) card in the Republic of Ireland, or for Northern Ireland patients, registered for NHS primary care services and registered with and/or regularly attending the practice for a minimum of 12 months). Each recruited GP practice will also display a patient recruitment poster in their practice waiting areas. Posters will direct patients to ask at reception if they are interested in taking part in the study.

The GP Practice Manager (or equivalent) will screen patient records facilitated and supported by the research nurses. Each practice will identify and filter potentially eligible participants via patient records. This will be done in batches depending upon the size of the practice list. Patients will be screened on the basis of the inclusion/exclusion criteria as specified in the protocol. A screening log will be provided to practices to record screening and recruitment activity, including the reason(s) for not being enrolled on the study. The screening log will be kept securely at the practice and no identifying data will leave the practice.

Intervention delivery: The intervention (video) will be delivered to recruited GPs allocated to the intervention arm using the 'Riverside' software programme. This software programme allows electronic, multimedia material to be delivered to healthcare professionals and students. GPs will be provided with a single generic username and password that will allow them to access the video on a secure online server. Prior to the commencement of the study, all participating GPs will be provided with instructions from the researcher on how to access the video. The researcher will be fully contactable during the study to answer any questions or queries that participating GPs may have about accessing the video.

Once consented, patients recruited by the GP practices allocated to the intervention arm will be asked to attend two appointments (telephone or online consultations where a face-to-face consultation is not possible) at a time convenient to them to have their medicines reviewed by a GP in addition to their usual care. Patients recruited by the GP practices allocated to the control arm will continue to receive usual care.

Data will be collected from recruited GPs, recruited patients and practice records. Recruited patients will be asked to complete a number of questionnaires relating to their general well-being and use of the health service (e.g. hospital admissions) at baseline, six months and nine months post-initial medication review in the intervention arm and the equivalent time points in the control arm. The follow up time points for the control arm will be based on the average length of time from the completion of baseline data collection to six and nine months post initial medication review in the intervention arm. Patient data (including medical history, clinical conditions, biochemical data (i.e. test results) and prescribed medications) will also be collected from GP records at baseline, six months and nine months by a Research Nurse from the Northern Ireland Clinical Research Network (NICRN Primary Care) or Trinity College Dublin (TCD).

At the end of the intervention, interviews will be conducted with up to 10 GPs and six members of practice staff (i.e. those involved in implementing the intervention within each practice) respectively in the six intervention arm practices. GPs will be asked about their views on the support provided by the research team; the intervention package (and supporting materials); study procedures (e.g. screening, recruitment, etc.), while practice staff will be asked about their views on the study procedures (e.g. screening, recruitment, etc.) and acceptability of the intervention. Patients from the six intervention group practices will be asked to complete a feedback questionnaire after the delivery of the intervention (i.e. after completion of their final follow-up questionnaires). Patients will be asked about their views on the study procedures (e.g. completing questionnaires, recruitment etc.) and acceptability of the intervention.

Who is funding the study: HSC R&D Division Cross-border Healthcare Intervention Trials in Ireland Network (CHITIN), UK and Ireland

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥70 years
* Patients must be receiving four or more regular medicines
* Patients must be resident in the community
* Patients must be in receipt of a valid general medical services (GMS) card in the Republic of Ireland, or in the case of Northern Ireland patients, registered for NHS primary care services
* Patients must be registered with and/or regularly attending the practice for a minimum of 12 months

Exclusion Criteria:

* Care home residents
* Patients who are cognitively impaired
* Patients with a terminal illness
* Involved in other Investigational Medicinal Product (IMP) or medicines management studies

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The number of patients contacted and recruited | Through study completion, an average of 1 year
The number of GP practices contacted and recruited | Through study completion, an average of 1 year
The retention rate of patients | Through study completion, an average of 1 year
  The number of patients retained over the study period
The retention rate of GP practices | Through study completion, an average of 1 year
  The number of GP practices retained over the study period
Medication appropriateness | Baseline
  Assessed using STOPP/START criteria
Medication appropriateness | Six months' post-initial medication review in the intervention arm and the equivalent time points in the control arm
  Assessed using STOPP/START criteria
Medication appropriateness | Nine months' post-initial medication review in the intervention arm and the equivalent time points in the control arm
  Assessed using STOPP/START criteria

SECONDARY OUTCOMES:
The number of video view counts per GP participant for the online video | Through study completion, an average of 1 year
  The number of times the GPs watched the online video; taken from the hosting website
The numbers of appointments scheduled | Through study completion, an average of 1 year
  Collected on study-specific data collection forms
The number of medication review appointments attended (first and second reviews) | Through study completion, an average of 1 year
  Collected on study-specific data collection forms
The length of the medication reviews | Through study completion, an average of 1 year
  The length of the medication reviews will be based on audio-recordings of a selection of patient medication reviews
The number of scheduled weekly meetings within each practice at which explicit plans were made to recall patients for medication reviews | Through study completion, an average of 1 year
  Recorded on GP practice staff data collection form
The number of prompts made by reception staff | Through study completion, an average of 1 year
  The number of prompts made by reception staff will be recorded on a GP practice staff data collection form
The resource use and associated costs of the intervention | Baseline, six months' post-initial medication review in the intervention arm and the equivalent time points in the control arm and nine months' post-initial medication review in the intervention arm and the equivalent time points in the control arm
Participant health and social care service use | Baseline, six months' post-initial medication review in the intervention arm and the equivalent time points in the control arm and 12 months' post--initial medication review in the intervention arm and the equivalent time points in the control arm
  As reported in GP notes and compared with self-reported health service use
Health-related quality of life | Baseline, six months' post-initial medication review in the intervention arm and the equivalent time points in the control arm and nine months' post-initial medication review in the intervention arm and the equivalent time points in the control arm
  Measured using the EQ-5D-5L
Medication-Related Burden Quality of Life | Baseline, six months' post-initial medication review in the intervention arm and the equivalent time points in the control arm and nine months' post-initial medication review in the intervention arm and the equivalent time points in the control arm
  Measured using the Medication-Related Burden Quality of Life (MRB-QoL) tool
Estimates of effect size between groups, cluster size and intraclass correlation coefficients (ICCs) | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Carmel Hughes, PhD, Principal Investigator — Queen's University, Belfast
Locations (2):
- Trinity College Dublin, Dublin, Ireland
- Queen's University Belfast, Belfast, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The current data sharing plans for this study are unknown and will be available at a later date

REFERENCES:
- [Background] Cadogan CA, Ryan C, Gormley GJ, Francis JJ, Passmore P, Kerse N, Hughes CM. A feasibility study of a theory-based intervention to improve appropriate polypharmacy for older people in primary care. Pilot Feasibility Stud. 2017 Jul 20;4:23. doi: 10.1186/s40814-017-0166-3. eCollection 2018. PMID 28748106
- [Background] Cadogan CA, Ryan C, Francis JJ, Gormley GJ, Passmore P, Kerse N, Hughes CM. Development of an intervention to improve appropriate polypharmacy in older people in primary care using a theory-based method. BMC Health Serv Res. 2016 Nov 16;16(1):661. doi: 10.1186/s12913-016-1907-3. PMID 27852287
- [Background] Rankin A, Cadogan CA, Barry HE, Gardner E, Agus A, Molloy GJ, Gorman A, Ryan C, Leathem C, Maxwell M, Gormley GJ, Ferrett A, McCarthy P, Fahey T, Hughes CM; PolyPrime team. An external pilot cluster randomised controlled trial of a theory-based intervention to improve appropriate polypharmacy in older people in primary care (PolyPrime): study protocol. Pilot Feasibility Stud. 2021 Mar 19;7(1):77. doi: 10.1186/s40814-021-00822-2. PMID 33741071
- [Background] Rankin A, Molloy GJ, Cadogan CA, Barry HE, Gorman A, Ryan C, Ferrett A, McCarthy P, Gormley GJ, Fahey T, Hughes CM; PolyPrime team. Protocol for a process evaluation of an external pilot cluster randomised controlled trial of a theory-based intervention to improve appropriate polypharmacy in older people in primary care: the PolyPrime study. Trials. 2021 Jul 14;22(1):449. doi: 10.1186/s13063-021-05410-6. PMID 34261527
- [Derived] Rankin A, Gorman A, Cole J, Cadogan CA, Barry HE, Agus A, Logan D, McDowell C, Molloy GJ, Ryan C, Leathem C, Maxwell M, Brennan C, Gormley GJ, Ferrett A, McCarthy P, Fahey T, Hughes CM; PolyPrime team. An external pilot cluster randomised controlled trial of a theory-based intervention to improve appropriate polypharmacy in older people in primary care (PolyPrime). Pilot Feasibility Stud. 2022 Sep 10;8(1):203. doi: 10.1186/s40814-022-01161-6. PMID 36088445